CLINICAL TRIAL: NCT05414929
Title: Prévention du Cancer du Col de l'UTÉrus Par dépistage d'Une Infection Partageable Sexuellement
Brief Title: Acceptability of HPV Self-sampling Among Canadian Women Aged 21 to 65
Acronym: CUTE-IPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Josianne Pare, Professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022-4535
Record Dates: First submitted 2022-03-10; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: HPV Infection; Cervical Cancer Screening
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV self-sampling group (Experimental)
  Interventions: Diagnostic Test: HPV self-sampling

INTERVENTIONS:
Diagnostic Test: HPV self-sampling — HPV self-sampling (Cobas Uniswab)

SUMMARY:
We propose a cross-sectional study to explore the acceptability and feasibility of HPV self-sampling among Quebec women. The study will invite eligible women to self-sample for HPV at home. The HPV risk factors of patients included in the study will be taken into consideration (vaccination, smoking, number of partners, date of last screening, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Speak and understand French without help

  * Have internet access (for completing forms)
  * Have a mailing address

Exclusion Criteria:

* Known positive HPV status • Have already had a hysterectomy

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the acceptability of HPV self-sampling by patients | 2 months following recruitment
  percentage of patients who prefer HPV testing to traditional cytology

SECONDARY OUTCOMES:
Evaluate the percentage of samples collected correctly by patients | 2 months following recruitment
Evaluate the return rate of mailed kits | 2 months following recruitment
Calculate the HPV positivity rate in a population sample | 2 months following recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Ruel-Laliberte J, Jacob-Wagner M, Bestman-Smith J, Pare J. Acceptability and Preferences of Dry HR HPV Self-Sampling Mailed Kits Among Canadian Women: A Cross-Sectional Study. J Obstet Gynaecol Can. 2023 Apr;45(4):261-266. doi: 10.1016/j.jogc.2023.02.012. Epub 2023 Mar 3. PMID 36870436